CLINICAL TRIAL: NCT06345430
Title: Clinical and Functional Effects of Wearable Technological Device Applied to Patients with Chronic Pain
Brief Title: Wearable Technological Device Applied to Patients with Chronic Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Ozlem Ulger, Professor, Hacettepe University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2023-14
Record Dates: First submitted 2023-11-16; First posted 2024-04-03 (Actual); Last update posted 2025-01-20 (Actual); Status verified 2025-01

CONDITIONS: Neck Pain; Low Back Pain; Chronic Pain; Musculoskeletal Pain
MeSH Terms: conditions — Neck Pain; Low Back Pain; Chronic Pain; Musculoskeletal Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Exopulse Molli Suit Interventipn (Experimental): After initial evaluations, patients received a single session for 1 hour. Exopulse Mollii Suit will be applied. The stimulation level of the electrodes will be determined by the automatically by the system in accordance with the level of pain they indicate for their parts, individually tailored to the person.
  will be created. Patients will wear the Exopulse Mollii Suit, which is suitable for their body size, Hacettepe University Physics They will dress in the room reserved for them at the Faculty of Treatment and Rehabilitation.
  Interventions: Device: Exopulse Molli-Suit (Wearable Technological Device)

INTERVENTIONS:
Device: Exopulse Molli-Suit (Wearable Technological Device) — After initial evaluations, patients will receive Exopulse Mollii Suit in a single session for 1 hour. The stimulation level of the electrodes will be automatically generated by the system in accordance with the pain level specified by the patients for their body parts before the application.

SUMMARY:
Within the scope of this research, a single session of Wearable Technological Device (Exopulse Molli-Suit) will be applied to patients with chronic back and neck pain. The results will be evaluated acutely, after 24 hours, after 1 week and after 1 month.

DETAILED DESCRIPTION:
After initial evaluations, patients received a single session for 1 hour. Exopulse Mollii Suit will be applied. The stimulation level of the electrodes will be determined by the automatically by the system in accordance with the level of pain they indicate for their parts, individually tailored to the person.

will be created. Patients will wear the Exopulse Mollii Suit, which is suitable for their body size, Hacettepe University Physics They will dress in the room allocated for them at the Faculty of Treatment and Rehabilitation. After each use The hygiene of Exopulse Mollii Suits has been evaluated at Hacettepe University Faculty of Physical Therapy and Rehabilitation in this will be provided with the help of a special device included in the scope. Initial assessments will be made immediately will be repeated three more times: after the intervention, 24 hours after the intervention and 4 weeks after the intervention.

All data will be collected face-to-face from patients using the instruments mentioned above.

ELIGIBILITY:
Inclusion Criteria:

* Being between the ages of 20-65
* Pain intensity should be at least 5 according to a numeric scale (low back pain and neck pain)
* no pain for at least 6 months (healthy people)

Exclusion Criteria:

* Malignant condition,
* People with systemic diseases such as neurological, psychological, cardiovascular, rheumatologic diseases and loss of function due to these diseases,
* History of previous surgery on the spine and upper extremities, including the cervical and lumbar region,
* Fractures in the spine and upper extremities, including the cervical and lumbar region, with a history of inflammation,
* Acute infection,
* Attending another rehabilitation program,
* Refused to participate in the study and did not give written informed consent

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2023-12-18 (Actual); Primary Completion 2024-04-15 (Actual); Study Completion 2024-06-30 (Actual)

PRIMARY OUTCOMES:
Pain Severity | bBefore the intervention, immediately after the intervention, after 24 hours, after 1 week and up to 1 month after the intervention. 5 times
  Numeric Pain Scale will be used. On a 10 cm horizontal straight line (0: no pain, 10: most severe pain), the patient will be asked to mark the relevant place according to the severity of the pain. Using a ruler, the distance between point 0 and the marked place will be measured to determine the intensity of the pain.

SECONDARY OUTCOMES:
Sleep Qaulity | Before the intervention, after 24 hours, after 1 week and up to 1 month after the intervention. 4 times
  In this evaluation, the Pittsburg Sleep Quality Index, which was developed by Buysse et al. (Buysse et al., 1989), and validated and reliably validated in Turkish by Ağargün et al. will be used (Ağargün et al., 1996). The index is presented in the appendix.
Disability Level | Before the intervention, after 24 hours, after 1 week and up to 1 month after the intervention. 4 times
  Oswestry Disability Index will be used for individuals with low back pain and Neck Disability Index for individuals with neck pain. The Turkish validity and reliability of the Oswestry Disability Index developed by Fairbank et al. (Fairbank & Pynsent, 2000) was demonstrated by Yakut et al. (Yakut et al., 2004) (internal consistency coefficient: 0.91). The Turkish validity and reliability of the Neck Disability Index developed by Vernon and Mior (Vernon & Mior, 1991) was demonstrated by Aslan et al. (Aslan et al., 2008) (internal consistency coefficient: 0.97).
Repetitive Reach Test | Before the intervention, after 24 hours, after 1 week and up to 1 month after the intervention. 4 times
  This test assesses the speed and coordination of the upper extremity in repetitive tasks. The time spent transferring 30 marbles (14 diameters) between two bowls placed at a distance determined by the arm opening is recorded in the sitting position. This test consists of four different subtasks, two-sided for the two upper extremities (right hand-left to the right, left hand-left to the right, right hand-right to the left, left hand-right to the left). Test-retest reliability in healthy subjects is weak
Body Composition Analysis | before intervention, 1 times
  Body Mass Index (BMI), muscular and fat body weights will be assessed with the TANITA BC420SMA (Tanita Corp, Tokyo, Japan). TANITA is a medically approved and reliable measuring device. It determines body composition by utilizing changes in bioelectric resistance (Jebb et al., 2000).
Lifting object overhead test | Before the intervention, after 24 hours, after 1 week and up to 1 month after the intervention. 4 times
  Lifitng object Overhead Test:This test is used to evaluate the functional strength of the upper extremity muscles. During the test, the participant takes the weight from a table 80 cm high and is asked to lift it up to the head five times within 90 seconds and return to the original position. It starts with the lightest weight determined and progresses step by step towards the heaviest. Initial and maximum weight were 10-60 kg and 6-30 kg in males and females, respectively. Increases are made in 4-5 kg (Gross & Battié, 2002). The criteria for termination of the test are reaching maximum weight, pain, or the individual's desire to terminate. Test-retest reliability in healthy subjects is high
Sustained Overhead Work Test | Before the intervention, after 24 hours, after 1 week and up to 1 month after the intervention. 4 times
  This test assesses postural tolerance capacity. The test is performed in the standing position with 1 kg cuff weights tied to the participant's arms. He was asked to manipulate the nuts and bolts as long as he can with the arms at forehead height and the time is recorded.
back performance test | Before the intervention, after 24 hours, after 1 week and up to 1 month after the intervention. 4 times
  evaluates the effectiveness of each activity that includes 5 different activities (socks test, gathering test, righting test, fingertip-floor test, carrying test). The Back Performance Scale test is scored between 0-15 points. An increase in score indicates a poor result

CONTACTS AND LOCATIONS:
Overall Officials: Özlem Ö Ülger, Proff, Study Director — Hacettepe Üniversity
Locations (1):
- Yasemin Özel Aslıyüce, Yenimahalle, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No